CLINICAL TRIAL: NCT02177474
Title: Randomized Controlled Trial of a Telephone Based Peer Support Intervention to Reduce Depressive Symptoms and Improve Social Support in Women With Coronary Heart Disease (CHD)
Brief Title: Effects of a Telephone Based Peer Support to Reduce Depressive Symptoms and Improve Social Support in Women With CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Kaufmännische Krankenkasse (KKH) (health insurance company) (Unknown)
Responsible Party: Principal Investigator, Christoph Herrmann-Lingen, Prof. Dr., University of Göttingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Frauenherz - 284; Frauenherz-Studie-284 (Other: IFS gGmbH)
Record Dates: First submitted 2014-06-19; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Depressive Symptoms; Low Perceived Social Support; Coronary Heart Disease
Keywords: depressive symptoms; perceived social support; coronary heart disease; peer support; women
MeSH Terms: conditions — Depression; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone based peer support (Experimental): The telephone based peer support was delivered by 11 women with chd aged 54 to 73 years, living all over Germany. Participants could call according to their needs during scheduled times on workdays.
  Interventions: Behavioral: Telephone based peer support
- Waitlist Group (Other): Waitlist condition with delayed telephone based peer support starting at 5 months
  Interventions: Behavioral: Telephone based peer support

INTERVENTIONS:
Behavioral: Telephone based peer support

SUMMARY:
In a randomized controlled trial the investigators intended to evaluate the effect of a telephone based peer support intervention on depressed or anxious women with coronary heart disease (CHD). The investigators intended to include 198 depressed or anxious women aged over 18 years with CHD. Participants were randomized to intervention (IG) or waiting list (WL). IG was offered immediate telephone-based contact to peer counselors while WL received the offer with a 6-month delay. All participants got at least one telephone call by a clinical psychologist (study information, feedback about the individual level of distress, proposal to get help). Main outcome variables were depressive symptoms (PHQ-9) and perceived social support (F-SozU K-14). In an additional quasi-experimental trial, the investigators included 11 peer counselors and 11 matched controls not taking part in the intervention. Main outcome variables were mood states (POMS) and perceived social support (F-SozU K-14).

ELIGIBILITY:
Inclusion Criteria:

* coronary heart disease
* depressive symptoms (HADS >7)
* insurants of former Kaufmännische Krankenkasse (KKH)-Allianz
* German speaking
* at least 18 years old
* written informed consent

Exclusion Criteria:

* hardness of hearing
* severe somatic illness
* current severe depressive episode or current suicidal tendency
* severe mental illness (dementia, psychosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change of Depressive Symptoms measured by PHQ-9 from baseline to 5 month | Baseline (T1), after 5 month (T2), after 11 month (T3)
  PHQ-9: Patient Health Questionnaire - Depression Scale
Change of perceived social support measured by F-SozU K-14 from baseline to 6 month | Baseline (T0), 5 month after T1 (T2), after 11 month (T3)
  F-SozU K-14: Fragebogen zur sozialen Unterstützung (Social Support Questionnaire)

SECONDARY OUTCOMES:
Change of Symptoms of anxiety measured by HADS-A from baseline to 5 month | Baseline (T1), after 5 month (T2), after 11 month (T3)
  HADS-A: Hospital Anxiety and Depression Scale - Anxiety Scale
Change of Self efficacy measured by SWE from baseline to 5 month | Baseline (T1), after 5 month (T2), after 11 month (T3)
  SWE: Fragebogen zur Allgemeinen Selbstwirksamkeitserwartung (Perceived self efficacy)
Change of Quality of life measured by WHOQOL-BREF from baseline to 5 month | Baseline (T1), after 5 month (T2), after 11 month (T3)
  WHOQOL-BREF: The World Health Organization Quality of Life-BREF

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Herrmann-Lingen, Prof. Dr., Study Director — University of Goettingen, Department of Psychosomatik Medicine and Psychotherapy
Locations (1):
- Department of Psychosomatic Medicine and Psychotherapy, Univ. of Göttingen, Göttingen, Germany